CLINICAL TRIAL: NCT02974673
Title: Ejaculation of Spinal Cord Patient: Pilot Study of Ejaculatory Dyssynergia by Electronic Microsensors of Sphincters
Brief Title: Pilot Study of Ejaculatory Dyssynergia by Electronic Microsensors of Sphincters
Acronym: EDGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-P0052; 2016-A01441-50 (Other: ANSM)
Record Dates: First submitted 2016-11-07; First posted 2016-11-28 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Spinal Cord Diseases; Disorder of Ejaculation
Keywords: Spinal Cord Injury; Genito sexuals disorders; Ejaculatory test
MeSH Terms: conditions — Spinal Cord Diseases; Ejaculatory Dysfunction; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ejaculatory test (Experimental): Measures of sphincter pressures during ejaculation
  Interventions: Procedure: Ejaculatory test

INTERVENTIONS:
Procedure: Ejaculatory test — Measures of sphincter pressures during ejaculation will be registered using a sensor introduced in the urethra on patient with spinal cord injury.

SUMMARY:
The objective of this research is to study the sphincter activity during ejaculation in patients with spinal cord injury in order to detect an ejaculatory dyssynergia. For this purpose, using a catheter the protocol plans to measure the sphincter pressures during ejaculation. Moreover, cardiovascular parameters will be measured continuously during the ejaculatory test.

ELIGIBILITY:
Inclusion Criteria:

* Patients evaluated by ejaculatory test during their usual care
* Men with spinal cord injury between 18 and 65 years old
* Patients who have given their informed consent
* Patients with social insurance affiliation

Exclusion Criteria:

* Minors
* Patients with justice protection
* Patients over 65 years old

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Sphincter urethral pressure measured by electronic microsensors to asses ejaculatory dyssynergia | at inclusion
  The presence of an ejaculatory dyssynergia will be certify by analysis of sphincter urethral pressure curves registered by microsensors during ejaculation

SECONDARY OUTCOMES:
Determination of type of ejaculation by bladder catheterization | at inclusion
  The type of ejaculation ( antegrade, retrograde or mixed) will be determined by searching sperm in urines due to a bladder catheterization after ejaculation
Sphincter urethral pressure to asses type of ejaculatory dyssynergia | at inclusion
  The type of ejaculatory dyssynergia will be determined by analysis of sphincter urethral pressures curves during ejaculation
American Spinal Injury Association score | at inclusion
  The neurological examination will be done by measuring the American Spinal Injury Association score, the international standard for evaluation of spinal cord injury
Frequency of ejaculation after stimulation | at inclusion
  The stimulation parameters will be measured during vibro massage
Amplitude of ejaculation after stimulation | at inclusion
  The stimulation parameters will be measured during vibro massage

CONTACTS AND LOCATIONS:
Overall Officials: Jean Gabriel Previnaire, MD, Study Director — Centre Calvé - Berck sur mer; Jean Marc Soler, MD, Principal Investigator — Center Bouffard Vercelli - Cerbère
Locations (2):
- France (2):
  - Centre Calvé, Berck
  - Centre Bouffard Vercelli, Cervera de la Marenda

IPD SHARING:
Plan to Share IPD: No